CLINICAL TRIAL: NCT05210712
Title: Respiratory Rate Validation Study - RS001.2 Respiree Cardio-Respiratory Monitor
Status: Completed | Type: Observational
Sponsor: Respiree Pte Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-462
Record Dates: First submitted 2022-01-12; First posted 2022-01-27 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-01

CONDITIONS: A Minimum of 30 Adults, Ages 18 Years and Older

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: RS001.2 Respiree Cardio-Respiratory Monitor — The RS001.2 Respiree Cardio-Respiratory Monitor is intended as a noninvasive multiparameter monitor on the adult population

SUMMARY:
The purpose of this study is to conduct a Respiratory Rate accuracy validation comparing the RS001.2 Respiree Cardio-Respiratory Monitor to the Reference, an FDA cleared End Tidal Carbon Dioxide monitor (GE Datex-Ohmeda).

DETAILED DESCRIPTION:
After IRB approval, a minimum of 30 volunteer test subjects will be enrolled for the final validation study population. A maximum of 60 subjects will be enrolled. All subjects will be 18 or older and selected to represent a range of body types including small, average, muscular, and large with a range of BMI's.

Each subject will be connected to a commonly used End Tidal Carbon Dioxide monitor (GE Datex-Ohmeda) and the RS001.2 Respiree Cardio-Respiratory Monitor. The end tidal carbon dioxide (EtCO2) monitor will determine performance of respiratory rate metrics (Reference). Each subject will be instrumented with a mouthpiece or nasal cannula that allows for measurement of the EtCO2. Subjects will also be connected to a 3-lead ECG and pulse oximeter in order to monitor the subject's vital signs for safety purposes.

Subjects will be seated for the study. A range of stable respiratory rates will be elicited from each volunteer test subject. After a baseline data set at the subject natural respiratory rate, the rates will be approximately 5, 10, 15, 20, 25, 30, 35, 40, 45, and 50 breaths per minute; with some natural variation from these exact numbers and tailored to the subject's capabilities. A paced breathing app will be used. It is expected that some of the subjects may not be able to be evaluated over the entire range as some subjects may not be able to breathe at the lower and higher respiratory rates. In this case, additional data may be recorded at the baseline range and other ranges that are comfortable for the subject. Once stable breathing at specified rate is achieved data will be collected for one to three minutes per respiratory rate plateau. Between plateaus, the subjects using a mouthpiece are allowed to take the mouthpiece out and relax.

The respiratory rate will be measured simultaneously with the Reference and the Device Under Test. During the stable plateaus at each level, the data will be averaged in approximately 60 second intervals. For final validation, the Reference EtCO2 waveform will be scored by counting the respiratory peaks per minute. The Accuracy root-mean-square (Arms) will be the basis for evaluation and acceptance.

To 'Pass' this test the RS001.2 Respiree Cardio-Respiratory Monitor (Device Under Test) must demonstrate an Accuracy root-mean-square (Arms) of ≤3 breaths per minute when compared to the Reference EtCO2 monitor.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have the ability to understand and provide written informed consent
* Subject must be ≥18 years of age
* Subject must be willing and able to comply with study procedures and duration
* Male or female of any race
* Baseline SpO2 ≥85%
* At least 3 subjects (10% of a total 30 subjects) will have a history of smoking

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

* Subjects who refuse or are unable to provide to sign an informed written consent for study
* Subject is evaluated by the Investigator and found to be medically unsuitable for participation in this study
* Compromised circulation, injury, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. Tattoo in the optical path which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the particular sites utilized.)
* Subjects with known respiratory conditions such as:

  * uncontrolled / severe asthma,
  * flu,
  * pneumonia / bronchitis,
  * shortness of breath / respiratory distress,
  * respiratory or lung surgery,
  * Severe COPD
* Subjects with self-reported heart or cardiovascular conditions such as:

  * high blood pressure: systolic >160 mmHg or diastolic >100 mmHg on 3 consecutive readings (reviewed during health screen)
  * have had cardiovascular surgery
  * chest pain (angina)
  * heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia (occasional PVCs is acceptable, less than two a minute)
  * previous heart attack
  * blocked artery
  * unexplained shortness of breath
  * congestive heart failure (CHF)
  * history of stroke
  * transient ischemic attack
  * carotid artery disease
  * myocardial ischemia
  * myocardial infarction
  * cardiomyopathy
* Self-reported health conditions as identified in the Health Assessment Form

  * uncontrolled thyroid disease,
  * kidney disease / chronic renal impairment,
  * history of seizures (except childhood febrile seizures),
  * epilepsy,
  * history of unexplained syncope,
  * recent history of frequent migraine headaches,
  * recent head injury within the last 2 months,
  * Cancer / chemotherapy
* Subjects with severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, or other medical sensors (self-reported)
* Other known health condition, should be considered upon disclosure in health assessment form

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will include a minimum of 30 healthy competent adults, ages 18 years and older. A maximum of 60 subjects will be enrolled.
  The subject selection will be a mix of males and females with small to large physiques. An attempt will be made to enroll a variety of skin tones. The goal is to include a range of skin pigmentations, including at least 5 darkly pigmented subjects or 15% of the subject pool, whichever is larger.
  The subjects must understand the study and consent to participate by signing the Informed Consent Form. Subject enrollment and participation in this clinical study is based on meeting the inclusion criteria and none of the exclusion criteria, a satisfactory health screen, and the subject and data demographics needed for the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Accuracy of the device to Reference | 1 to 3 minutes at a given level
  The primary objective of this study is to compare the accuracy of the device under test for the measurement of respiratory rate to the Reference, which is an End Tidal Carbon Dioxide Monitor (EtCO2). For final validation, the EtCO2 waveform will be scored by counting the respiratory peaks per minute.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinimark, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No